CLINICAL TRIAL: NCT04054076
Title: 10 Years Follow-up of Gait Characteristics, Plantar Pressure, Kinetics and Kinematics in a Cohort of Patients Diagnosed With Diabetes
Brief Title: 10 Years Follow-up Study of Plantar Pressure, Kinetics and Kinematics in a Cohort of Patients Diagnosed With Diabetes
Acronym: Diab10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Ulla Hellstrand Tang, Principal Investigator, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SU-896191
Record Dates: First submitted 2019-07-25; First posted 2019-08-13 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Diabetes; Diabetic Foot; Plantar Ulcer; Neuropathy; Gait Disorder, Sensorimotor; Motor Neuropathy; Foot Deformities; Foot Ulcer
Keywords: orthotics; kinematics; kinetics
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Foot Ulcer; Gait Disorders, Neurologic; Neuritis; Foot Deformities

STUDY DESIGN:
Intervention Model Description: This study is a 10 year follow-up of an original randomized clinical trial (RCT) study (n= 114 patients) with type 1 and type 2 diabetes. The participants were referred to the department of Prosthetics & Orthotics (DPO) at Sahlgrenska University Hospital and were randomised to: 1) use prefabricated insoles, 2) soft custom-made insoles or 3) hard custom-made insoles. The groups were followed 2 years with follow-ups every 6 months. Data regarding plantar pressure, gait characteristics, kinetics and kinematics and presence of risk factors will be collected 10 years after inclusions. Comparisons will be made with a group of patients with diabetes being first times visitors to the Department of Prosthetics & Orthotics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prefabricated insoles (Experimental): Prefabricated insoles with support in medial arch and metatarsal pad. A 2 mm top layer of cushioned material.
  Interventions: Device: Prefabricated insoles
- Custom-made insoles soft (Experimental): Custom-made insoles formed over an individual cast positive. 35 shore of hardness in material Ethyl Vinyl Acetate.
  Interventions: Device: Soft custom-made insoles
- Custom-made hard (Experimental): Custom-made insoles formed over an individual cast positive. 55 shore of hardness in material Ethyl Vinyl Acetate.
  Interventions: Device: Hard custom-made insoles
- Control group (No Intervention): No intervention with therapeutic insoles and/or shoes.

INTERVENTIONS:
Device: Prefabricated insoles — The participants received prefabricated insoles
  Arms: Prefabricated insoles
Device: Soft custom-made insoles — The participants received soft custom-made insoles
  Arms: Custom-made insoles soft
Device: Hard custom-made insoles — The participants received hard custom-made insoles
  Arms: Custom-made hard

SUMMARY:
A combination of diabetes and neuropathy can cause an altered gait, increased tissue stiffness, limited joint mobility, muscle weakness, foot deformities, thus leading to excessive plantar pressure. The presence of an increased plantar pressure and the loss of sensation is a serious risk factor in the risk of development of diabetic foot ulcers (DFU). Therefore, appropriate shoes and insoles are recommended to redistribute high peak pressure (PP) and reduce pressure time integral (PTI) . Shoe modifications and insoles, when used, is effective to prevent the recurrence of plantar ulcer.

The primary aim of the study was to: explore gait characteristics, kinetics and kinematics in a cohort of patients diagnosed with diabetes, with and without neuropathy, assigned to use different types of insoles. The second aim was to assess the relation between gait characteristics, kinetics and kinematics to high plantar PP and PTI. The third aim was to compare gait characteristics, kinetics and kinematics of patients with diabetes and healthy controls.

DETAILED DESCRIPTION:
A combination of diabetes and neuropathy can cause an altered gait, increased tissue stiffness, limited joint mobility, muscle weakness, foot deformities, thus leading to excessive plantar pressure . The presence of an increased plantar pressure and the loss of sensation is a serious risk factor in the risk of development of diabetic foot ulcers (DFU). Therefore, appropriate shoes and insoles are recommended to redistribute high peak pressure (PP) and reduce pressure time integral (PTI). Shoe modifications and insoles, when used, is effective to prevent the recurrence of plantar ulcer.

Patients presenting with mild or absence of neuropathy have lower PP compared to those having more severe stages of neuropathy. However, these findings are not unambiguous. In a study patients walked in a standardize speed of 1.2 m/s, and it was only under the first metatarsal phalangeal joint that the group with neuropathy had higher PP compared to patients with diabetes without neuropathy. In the remaining parts of the foot sole, there was no difference. In a study comparing custom-made insoles and prefabricated insoles used in a walking shoe, a cohort of patients with no history of foot ulcers was studied and there were no differences in PP for the sub groups with and without neuropathy.

More knowledge is needed regarding risk factors such as neuropathy, gait deviation and differences in kinematics and kinetics in order to prevent the onset of the "first" plantar ulcer.

ELIGIBILITY:
Inclusion Criteria:

Intervention groups:

* To be a participant in the original RCT
* To be aged 18 years or more
* To walk without walking aid
* To understand the Swedish language
* No presence of foot ulcer

Exclusion Criteria:

* Presence of foot ulcers

Control group

* To be first-time visitors to the DPO
* To be aged 18 years or more
* To walk without walking aid
* To understand the Swedish language
* No presence of foot ulcer

Exclusion Criteria:

* Presence of foot ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Peak pressure | through study completion, an average of 1 year
  To compare the differences of peak pressure (kPa) in the four groups.
Pressure time integral | through study completion, an average of 1 year
  To compare the differences of pressure time integral (kPa*s) in the four groups.

SECONDARY OUTCOMES:
Moment at ankle-knee-and hip joint | through study completion, an average of 1 year
  To compare the differences of joint moment (Nm/kg) in the four groups.
Speed | through study completion, an average of 1 year
  To compare the differences of speed (m/s) in the four groups.
Cadence | through study completion, an average of 1 year
  To compare the differences of cadence (step/min) in the four groups.
Stance (percent of stand phase) | through study completion, an average of 1 year
  To compare the differences of stance phase (%) in the four groups.
Range of foot-knee and hip angles (minimum to maximum) | through study completion, an average of 1 year
  To compare the differences of maximum angle (degree) in the four groups
Walking distance of 5 minutes walking | through study completion, an average of 1 year
  To compare the differences of 5 minutes walking(m) distance in the four groups
Distribution of risk grade ( the risk to develop diabetic foot ulcers 1-4(1=no risk, 4=presence of foot ulcers) | through study completion, an average of 1 year
  To assess the distribution of risk grade (1-4) in the four groups
Relation of different types of insoles and risk factors to peak pressure | through study completion, an average of 1 year
  To assess the influence of different types of insoles and risk factors on high peak pressure (kPa)
Relation of different types of insoles and risk factors to pressure time integral | through study completion, an average of 1 year
  To assess the influence of different types of insoles and risk factors on pressure time integral (kPa*s)

OTHER OUTCOMES:
Health related quality of life | through study completion, an average of 1 year
  To assess the quality of life (SF-36 and EQ-5D-5L) in the different groups
Costs for the assistive devices | through study completion, an average of 1 year
  Calculation of costs (SEK and USD) for the assistive devices

CONTACTS AND LOCATIONS:
Overall Officials: Björn Stålgren, BSc, Study Director — Sahlgrenska University Hospital
Locations (1):
- Department of Prostetics & Orthotics, Gothenburg, Region Västragötaland, Sweden

IPD SHARING:
Plan to Share IPD: No